CLINICAL TRIAL: NCT00206739
Title: Intermittent Treatment With Sulfadoxine-pyrimethamine for Malaria Control in Infant: a Randomized, Double-blind, and Placebo-controlled Clinical Trial
Brief Title: Intermittent Treatment With Sulfadoxine-pyrimethamine for Malaria Control in Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bernhard Nocht Institute for Tropical Medicine (Other Government)
Collaborators: German Federal Ministry of Education and Research (Other Government); Deutscher Akademischer Austausch Dienst (Other); The Volkswagen Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01KA0202-K7.3; 01KA0202
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2005-09

CONDITIONS: Malaria; Anemia
Keywords: Malaria; Anemia; IPTi; Intermittent Preventive Treatment in Infants; Sulfadoxine-Pyrimethamine; Chemoprophylaxis; Ghana
MeSH Terms: conditions — Malaria; Anemia | interventions — Sulfadoxine; Pyrimethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sulfadoxine (12.5 mg)/Pyrimethamine (250 mg)

SUMMARY:
The purpose of this study is to assess the effectiveness of Intermittent Preventive Treatment in Infants (IPTi) with Sulfadoxine-Pyrimethamine to reduce the numbers of malaria attacks, episodes of anemia, and the overall morbidity and mortality

DETAILED DESCRIPTION:
In order to define the effectiveness of Intermittent Preventive Treatment in Infants (IPTi) with Sulfadoxine-Pyrimethamine, a novel principle of malaria intervention, the following parameters are evaluated: i) the level of protection from malaria attacks and episodes of anemia during the treatment period, ii) the level of protection from severe malaria during the treatment period, iii) the effect on malaria morbidity after sustaining treatment, iv) the decrease of overall morbidity and mortality, including the number of hospital admissions and visits of hospital outpatient departments v) the influence of the intervention on the development of drug resistances, vi) the impact of the intervention on the development of immunity, vii) the possible influence of the intervention on sub-clinical organ dysfunction due to chronic Plasmodium falciparum infection. Parts of the study are performed in collaboration with the Laboratory of Research, Hospital Albert Schweitzer, Lambaréné, Gabon and the School of Medicine and Health Sciences, University of Development Studies, Tamale, Ghana

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by parent/guardian (written or oral)
* Permanent residentship in the study area
* Age of 3 months +/-4 weeks

Exclusion Criteria:

* Hypersensitivity to sulfonamides or pyrimethamine (skin rashes, evidence of hemolysis including dark urine and/or purpura, presumptive signs of bone marrow depression such as sore throat and/or mouth ulcers)
* Other severe adverse events related to pyrimethamine-sulfadoxine application
* Signs of severe hepatic or renal dysfunction not due to malaria
* Other reasons after decision of the study physician

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1070 (Actual)
Dates: Start 2003-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
• Efficacy of an extended intermittent treatment with sulfadoxine-pyrimethamine for the control of clinical malaria and anemia (proportion and rates of children with one or more episodes of malaria or anemia in the age of 3 to 21 months of life)
• Determination of the rate of clinical malaria and anemia after suspending an extended intermittent treatment for analysis of possible rebound effects
• Evaluation of safety and adverse effects of the administration of single doses of sulfadoxine-pyrimethamine in infants and children

SECONDARY OUTCOMES:
• Rate and time points of hospitalizations with anemia, malaria or other diseases
• Rate and time points of severe anemia episodes
• Proportion and rates of children with one or more episodes of malaria or anemia in the age of 3 to 12 months of life
• Antibody responses against parasite antigens
• Multiplicity of P. falciparum infections
• Proportion of P. falciparum isolates with SP resistance
• Influence of host genetic variants on the rate of P. falciparum infections

CONTACTS AND LOCATIONS:
Overall Officials: Ohene Adjei, Prof. Dr., Principal Investigator — Kumasi Centre for Collaborative Research in Tropical Medicine; Jürgen May, PD Dr., Study Director — Bernhard Nocht Institute for Tropical Medicine Hamburg, Infection Epidemiology
Locations (1):
- Kumasi Centre for Collaborative Research in Tropical Medicine, Kumasi, Ashanti Region, Ghana

REFERENCES:
- [Background] Schellenberg D, Menendez C, Kahigwa E, Aponte J, Vidal J, Tanner M, Mshinda H, Alonso P. Intermittent treatment for malaria and anaemia control at time of routine vaccinations in Tanzanian infants: a randomised, placebo-controlled trial. Lancet. 2001 May 12;357(9267):1471-7. doi: 10.1016/S0140-6736(00)04643-2. PMID 11377597
- [Background] Menendez C, Kahigwa E, Hirt R, Vounatsou P, Aponte JJ, Font F, Acosta CJ, Schellenberg DM, Galindo CM, Kimario J, Urassa H, Brabin B, Smith TA, Kitua AY, Tanner M, Alonso PL. Randomised placebo-controlled trial of iron supplementation and malaria chemoprophylaxis for prevention of severe anaemia and malaria in Tanzanian infants. Lancet. 1997 Sep 20;350(9081):844-50. doi: 10.1016/S0140-6736(97)04229-3. PMID 9310602
- [Background] Massaga JJ, Kitua AY, Lemnge MM, Akida JA, Malle LN, Ronn AM, Theander TG, Bygbjerg IC. Effect of intermittent treatment with amodiaquine on anaemia and malarial fevers in infants in Tanzania: a randomised placebo-controlled trial. Lancet. 2003 May 31;361(9372):1853-60. doi: 10.1016/s0140-6736(03)13504-0. PMID 12788572
- [Background] Verhoef H, West CE, Nzyuko SM, de Vogel S, van der Valk R, Wanga MA, Kuijsten A, Veenemans J, Kok FJ. Intermittent administration of iron and sulfadoxine-pyrimethamine to control anaemia in Kenyan children: a randomised controlled trial. Lancet. 2002 Sep 21;360(9337):908-14. doi: 10.1016/S0140-6736(02)11027-0. PMID 12354473
- [Derived] May J, Adjei S, Busch W, Gabor JJ, Issifou S, Kobbe R, Kreuels B, Lell B, Schwarz NG, Adjei O, Kremsner PG, Grobusch MP. Therapeutic and prophylactic effect of intermittent preventive anti-malarial treatment in infants (IPTi) from Ghana and Gabon. Malar J. 2008 Oct 1;7:198. doi: 10.1186/1475-2875-7-198. PMID 18828899
- [Derived] Kobbe R, Adjei S, Kreuzberg C, Kreuels B, Thompson B, Thompson PA, Marks F, Busch W, Tosun M, Schreiber N, Opoku E, Adjei O, Meyer CG, May J. Malaria incidence and efficacy of intermittent preventive treatment in infants (IPTi). Malar J. 2007 Dec 9;6:163. doi: 10.1186/1475-2875-6-163. PMID 18067679
- See also: Homepage of the Kumasi Centre for Collaborative Research (study site) — http://www.kccr.de/kccr/